CLINICAL TRIAL: NCT06442384
Title: Fully Remote Randomized Controlled Trial Exploring the Role of Non-combustible Tobacco Products in the Context of a Nicotine Product Standard for Cigarettes
Brief Title: Remote Trial - Tobacco Product Standard (VLNC)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study determined to be not feasible at this time due to limited availability of study product and limited availability of study products in the marketplace.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023LS188
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Tobacco Use
Keywords: reducing nicotine cigarettes
MeSH Terms: conditions — Tobacco Use | interventions — Tobacco Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VLNC cigarettes plus access to tobacco and non-tobacco flavored e-cigarettes (Experimental): Smokers who meet eligibility criteria will enter 2 weeks of monitoring of usual brand smoking. Participants will then be randomly assigned to a 4-week intervention
  Interventions: Other: Tobacco and non-tobacco e-cigarettes
- VLNC cigarettes plus access to only tobacco flavored e-cigarettes (Experimental): Smokers who meet eligibility criteria will enter 2 weeks of monitoring of usual brand smoking. Participants will then be randomly assigned to a 4-week intervention
  Interventions: Other: Tobacco only e-cigarettes

INTERVENTIONS:
Other: Tobacco and non-tobacco e-cigarettes — Participants with no e-cigarette restrictions.
  Arms: VLNC cigarettes plus access to tobacco and non-tobacco flavored e-cigarettes
Other: Tobacco only e-cigarettes — Participants restricted to tobacco flavored e-cigarettes only.
  Arms: VLNC cigarettes plus access to only tobacco flavored e-cigarettes

SUMMARY:
The goal of this pilot project is to explore the feasibility of a real-world marketplace study design examining the effects of a reduced nicotine product standard for cigarettes on smoking in the context of a flavor restriction vs. no restriction on e-cigarettes in smokers switched to very low nicotine content cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* Self-report of daily smoking of at least 5 to 25 cigarettes for >3 months by self-report.
* Carbon monoxide indicative of regular smoking (CO > 6ppm) prior to randomization.
* Has regular access to a smartphone, tablet or computer with functioning camera and internet access for telehealth visits and surveys and to take photos of receipts.
* Lives in an area where VLN® cigarettes are being marketed (these locations may vary during the course of the study).

Exclusion Criteria:

* Unstable health conditions (any significant serious, unstable medical condition including, but not limited to, cardiovascular disease, liver or kidney disease, COPD, bronchitis, within the past 3 months, seizure disorder and cancer (cancer-free <5 years except some skin cancers can be within 5 years), or a COVID-19 positive test or COVID-19 symptoms in the last 14 days or as determined by the licensed medical professional at each site).
* Unstable mental health (to be determined by medical history, Patient Health Questionnaire-2 (Prime-MD) and GAD-2 after review by the licensed medical professional).
* Excessive drinking or problems with drinking or drugs-including marijuana (assessed by PI or licensed medical professional).
* Currently pregnant, breastfeeding or intending to become pregnant for the duration of the study or unwilling to agree to use adequate protection to avoid pregnancy.
* Taking exclusionary medications, unstable dosing of medications, or unstable control of symptoms for ongoing medical conditions (medications or conditions that would impact patient safety to be determined by the licensed medical professional).
* Recent experience with VLNC cigarettes (purchasing of the VLNC cigarettes in the past year)
* Household member enrolled in the study concurrently.
* Participated in prior research study during the past three months that would impact baseline smoking or response to study products.
* Inability to independently read and comprehend the consent form and follow other written study instructions, materials or measures or behavior indicating inability to fully participate in study procedures. Participants are required to complete the protocol at home independently and must show ability to comply with directions.
* Unstable living environment that would compromise the ability to sequester study products or complete study procedures.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Percent of participants that drop-out by 4 week visit | 4 weeks
  Percent of participants that drop-out by 4 week visit

SECONDARY OUTCOMES:
Change in mean cigarettes per day (CPD) | Baseline to 4 weeks
  Change in mean cigarettes per day (CPD) based on 7 day ITR data before visit 00 and week 4 visits
Number of participants experiencing smoke free days | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Masonic Cancer Center, Minneapolis, Minnesota, United States